CLINICAL TRIAL: NCT06433297
Title: Comparative Evaluation of Indirect and Direct Pulp Capping After Partial or Complete Caries Removal in Deeply Carious Mature Permanent Mandibular Molars With Moderate Pulpitis: A Randomized Clinical Trial
Brief Title: Comparative Evaluation of Indirect vs. Direct Pulp Capping in Deep Carious Mandibular Molars
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Soma Chanakya
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Indirect Pulp Capping; Reversible Pulpitis
Keywords: indirect pulp capping; selective caries removal; moderate pulpitis; direct pulp capping; deep caries; complete caries removal; mature permanent mandibular molars

STUDY DESIGN:
Who Masked: Participant
Masking Description: Considering the nature of intervention, masking of the operator will not be possible once he begins the caries removal. Patients will be unaware of the groups in which their allocation will take place. At the time of assessing data masking will be done by masking the entire crown of the tooth before evaluation by endodontist using Adobe Photoshop CS6.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Partial caries removal followed by Indirect pulp capping. (Experimental): Partial caries removal followed by Indirect pulp capping.
  Interventions: Procedure: INDIRECT AND DIRECT PULP CAPPING AFTER PARTIAL OR COMPLETE CARIES REMOVAL IN DEEPLY CARIOUS MATURE PERMANENT MANDIBULAR MOLARS WITH MODERATE PULPITIS
- Complete caries removal followed by Direct Pulp Capping (Active Comparator): Complete caries removal followed by Direct Pulp Capping
  Interventions: Procedure: INDIRECT AND DIRECT PULP CAPPING AFTER PARTIAL OR COMPLETE CARIES REMOVAL IN DEEPLY CARIOUS MATURE PERMANENT MANDIBULAR MOLARS WITH MODERATE PULPITIS

INTERVENTIONS:
Procedure: INDIRECT AND DIRECT PULP CAPPING AFTER PARTIAL OR COMPLETE CARIES REMOVAL IN DEEPLY CARIOUS MATURE PERMANENT MANDIBULAR MOLARS WITH MODERATE PULPITIS — After partial caries removal the cavity is disinfected, dried, and capped with a 2-3mm layer of MTA followed by a light-cured resin layer. The tooth is then definitively restored with composite.
  Following complete caries removal, any bleeding pulp will be controlled with sodium hypochlorite for up to 5 minutes. Exposed pulp will then be directly capped with a 2-3mm layer of MTA, followed by a light-cured resin layer and definitive composite restoration using an etch-and-rinse technique.

SUMMARY:
Aim: To compare the outcome of indirect and direct pulp capping after partial or complete caries removal in deeply carious mature mandibular permanent molars with clinical signs indicative of moderate pulpitis.

Objectives:

1. To evaluate the clinical and radiographic success of indirect pulp capping after partial caries removal in deeply carious mature mandibular permanent molars with clinical signs indicative of moderate pulpitis.
2. To evaluate the clinical and radiographic success of direct pulp capping after complete caries removal in deeply carious mature mandibular permanent molars with clinical signs indicative of moderate pulpitis.
3. To evaluate pain incidence and severity after indirect and direct pulp capping after partial and complete caries removal in deeply carious mature mandibular permanent molars with clinical signs indicative of moderate pulpitis.

DETAILED DESCRIPTION:
Vital pulp therapy has been traditionally recommended only in teeth with reversible pulpitis with no periapical pathologies or in teeth with either mechanical pulp exposure or recent traumatic exposure. Clinical symptoms such as characteristics, severity and intensity of pre-operative pain do not accurately talk about the status of the pulp inflammation and the depth of involvement. It has been demonstrated that there is no precise correlation between clinical symptoms and the histopathological status of the pulp, mainly in case of irreversible pulpitis, that might lead to a wrong diagnosis. Vitality tests such as cold test or electric pulp tests reveal only whether the pulp is responsive to respective stimuli or not. According to new Wolters pulpal clinical classification, Moderate pulpitis exhibit symptoms of prolonged reaction to cold, which can last for minutes, possibly percussion sensitive and spontaneous dull pain which corresponds to irreversible pulpitis. Vital pulp therapy is suggested to be the choice of treatment for such cases. It has been suggested that infection is often a cause of inflammation, an inflamed pulp should be able to heal if the source of infection is eliminated as in other body organs. Removal of trigger (i.e. caries) followed by application of biocompatible material which makes a good seal in a sterile environment has potential to allow for recovery and healing of the inflamed pulp tissue which is thought to be beyond recovery. Partial caries removal, which involves complete removal of carious dentine from the surrounding cavity walls, followed by the partial removal of infected dentin at the pulpal wall which reduce chances of pulp exposure followed by placement of medicament for Indirect pulp capping. Whereas during Complete caries removal, caries is completely removed from surrounding walls as well as on pulpal wall which increase the chances of pulp exposure followed by placement of medicament for Direct pulp capping procedure. Based on this premise, IPC can be considered as minimally invasive approach for the management of teeth with inflamed pulps in place of the conventional approach of direct pulp capping, partial pulpotomy or full pulpotomy in adults.

Research Question Does Indirect Pulp Capping have comparable outcome with Direct pulp capping after partial caries removal in deeply carious mature permanent molars with clinical signs indicative of moderate pulpitis? P (Population) - Deeply carious mature Permanent Mandibular molars with clinical signs indicative of moderate pulpitis I (Intervention) - Partial caries removal followed by Indirect pulp capping C (Comparison) - Complete caries removal followed by Direct pulp capping O (Outcome) - Assessment of clinical and radiographic success at 12 months follow up.

* To assess incidence and reduction in pain post operatively at every 24 hours till 1 week.

ELIGIBILITY:
Inclusion Criteria:

1. The patient should be ≥18 years of age.
2. Restorable mature permanent 1st and 2nd Mandibular molars with deep caries (reaching inner quarter of dentine)
3. Tooth should give positive response to pulp sensibility testing.
4. Clinical diagnosis of moderate pulpitis.
5. Radiographic finding of periapical index (PAI) score ≤2.
6. Healthy periodontium (probing pocket depth ≤3 mm and mobility within normal limit).
7. Pulp exposure after complete caries excavation.
8. No pulp exposure after incomplete caries excavation

Exclusion Criteria:

1. Teeth with immature roots.
2. Pulp exposure after incomplete caries excavation.
3. No pulp exposure after complete caries excavation.
4. Bleeding could not be controlled in 5 minutes.
5. Signs of pulpal necrosis, sinus tract, swelling, insufficient bleeding after pulp exposure.
6. History of analgesic intake in previous 1 week, or antibiotic intake in 1 month.
7. Internal/external resorption.
8. Contributory medical history (alcoholism, smokers, diabetic, hypertension, drug dependency, Heart or valve disease, hepatitis, herpes, immunodeficiency (HIV), infectious diseases, kidney or liver, migraine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2026-03-23 (Estimated); Study Completion 2026-03-23 (Estimated)

PRIMARY OUTCOMES:
Clinical Success Rate | 12 months
  No pain or discomfort. No tenderness to palpation or percussion. Normal mobility and probing pocket depth.
Radiographic success | 12 months
  No pathology on the radiograph.

SECONDARY OUTCOMES:
Pain reduction | Seven days
  Post operative pain To assess pain postoperatively at every 24 hours till 7 days using Visual analogue Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Dr, Sanjay Tewari, MDS, Study Director — PGIDS, Rohtak, Haryana, 124001
Locations (1):
- PGIDS, Rohtak, Rohtak, Haryana, India